CLINICAL TRIAL: NCT01381068
Title: Quantitative End Tidal CO2 Monitoring in the Delivery Room: Can we Prevent Hypo/Hypercapnia Upon Admission to the NICU?
Brief Title: Quantitative End Tidal CO2 Monitoring in the Delivery Room (DR)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neil Finer (Other)
Responsible Party: Sponsor-Investigator, Neil Finer, Professor Emeritus, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 090780
Record Dates: First submitted 2011-06-21; First posted 2011-06-27 (Estimated); Results first posted 2019-12-17 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-10

CONDITIONS: Delivery Room Resuscitation
Keywords: ventilation; end tidal carbon dioxide; hypercapnia; hypocapnia; positive pressure ventilation; neonates; delivery room resuscitation
MeSH Terms: conditions — Respiratory Aspiration; Hypercapnia; Hypocapnia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Monitored Arm (Experimental): The end tidal CO2 sensor is placed in the respiratory circuit and the monitor is visible to the resuscitation team. The resuscitation team is instructed to adjust ventilation to keep EtCO2 levels between 40-55.
  Interventions: Device: End tidal CO2 monitor
- Control Arm (Placebo Comparator): The end tidal CO2 sensor is placed in th respiratory circuit. The monitor is covered so the resuscitation team can not see the display. The resuscitation team is instructed to provide ventilation according to clinical judgment.
  Interventions: Device: End tidal CO2 monitor

INTERVENTIONS:
Device: End tidal CO2 monitor — The sensor is placed in the respiratory circuit in both arms of the trial but the display is visible to the resuscitation team in the monitored arm and is covered in the control arm. The end tidal CO2 data is collected in both arms.
  Other Names: NICO 2 Respiratory Profile Monitor (Respironics, Inc.)

SUMMARY:
This is a trial evaluating the use of an end tidal CO2 monitor during ventilation in the delivery room. The use of the monitor is compared with clinical assessment of ventilation. The hypothesis is that using the monitor would results in a decrease in the incidence of hypo- or hypercapnia on admission to the NICU.

ELIGIBILITY:
Inclusion Criteria:

* Need for ventilation in the delivery room

Exclusion Criteria:

* Tracheal suctioning for meconium
* Congenital Diaphragmatic Hernia
* Suspected hypoplasia of the lungs
* Oligohydramnios <28 weeks gestation or AFI<5
* Known or suspected airway anomaly
* Mother not speaking English or Spanish
* Refusal of consent

Max Age: 15 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2009-10 (Actual); Primary Completion 2011-05 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tina A Leone, MD, Principal Investigator — UCSD
Locations (1):
- UCSD Medical Center, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 50 participants were randomized however one participants randomization assignment was undocumented, so 49 participants are accounted for.
Period: Overall Study
Arm/Group | Monitored Arm | Control Arm
Started (one infant had an unassigned randomization and was not included) | 25 | 24
Completed | 24 | 24
Not Completed | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Population: 50 participants were randomized however one participants randomization assignment was undocumented and one participant died, so the results are being recorded for 48 subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | Monitored Arm | Control Arm | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Customized [Mean (Full Range); unit: weeks]
  Age ( Gestational Age , weeks and range | 28.9 [24.6 to 35.3] | 29.3 [24.9 to 35.1] | 29.2 [24.6 to 35.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 12 | 30
  Male | 6 | 12 | 18
Antenatal Steroids [Count of Participants; unit: Participants] | 23 | 23 | 46
Mode of Delivery - Cesarean Section [Count of Participants; unit: Participants] | 19 | 17 | 36
5 mim Apgar < 5 [Count of Participants; unit: Participants] | 0 | 1 | 1
Twin [Count of Participants; unit: Participants] | 7 | 4 | 11
DR Intubation [Count of Participants; unit: Participants] | 3 | 4 | 7
NICU Intubation [Count of Participants; unit: Participants] | 9 | 10 | 19
DR CPR [Count of Participants; unit: Participants] | 0 | 0 | 0
Cord PCO2 (mmHg) [Mean (Full Range); unit: mmHg] | 52 [37 to 83] | 50 [40 to 63] | 51 [37 to 83]
Rec'd Surfactant [Count of Participants; unit: Participants] | 12 | 13 | 25

OUTCOME MEASURES:

1. Primary Outcome: PCO2 Level Outside of Desired Range (40-60 mmHg)
Description: This outcome will be obtained from the first available blood gas after admission to the NICU.
Time Frame: Admission to NICU, approximately 1 hour of life
Measure: Number; unit: participants
Arm/Group | Monitored Arm | Control Arm
Number analyzed (Participants) | 24 | 24
participants | 9 | 8

2. Secondary Outcome: End Tidal CO2 Levels
Description: The EtCO2 levels from the last 5 breaths of the DR resuscitation will be averaged to determine this outcome.
Time Frame: At the conclusion of resuscitation, approximately 15 minutes of life.
Measure: Mean (Full Range); unit: mmHg
Arm/Group | Monitored Arm | Control Arm
Number analyzed (Participants) | 24 | 24
mmHg | 42.8 [29 to 59] | 44.3 [16 to 66]

3. Secondary Outcome: Duration of Ventilation
Description: The number of days on the ventilator during the entire hospital course will be counted for this outcome.
Time Frame: Duration of the hospital course, approximately 2-3 months
Measure: Mean (Full Range); unit: days
Arm/Group | Monitored Arm | Control Arm
Number analyzed (Participants) | 24 | 24
days | 1 [0 to 30] | 1.5 [0 to 38]

4. Secondary Outcome: Oxygen Use at 36 Weeks
Description: This outcome will be counted as yes if the infant is receiving oxygen at 36 weeks adjusted age.
Time Frame: Hospital course, approximately 2-3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Monitored Arm | Control Arm
Number analyzed (Participants) | 24 | 24
Participants | 3 | 2

5. Secondary Outcome: Incidence of Pneumothorax/Airleak
Description: This outcome will be counted as yes if any pneumothorax or airleak is noted on any chest xray during the hospitalization.
Time Frame: Hospital course, approximately 2-3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Monitored Arm | Control Arm
Number analyzed (Participants) | 24 | 24
Participants | 2 | 2

6. Secondary Outcome: Number of Patients Ventilated on NICU Admission
Description: At the time of NICU admission directly after the DR resuscitation the number of patients ventilated will be reported per group
Time Frame: On NICU admission, approximately 15 minutes of life
Population: Only 7 patients were ventilated on admission to the NICU- data not presented
Measure: Count of Participants; unit: Participants
Arm/Group | Monitored Arm | Control Arm
Number analyzed (Participants) | 24 | 24
Participants | 3 | 4

7. Secondary Outcome: Systemic Blood Flow - as Measured by Supervior Vena Cava (SVC) Flow
Description: An echocardiogram performed within the first 12 hours of life will measure supervior vena cava (SVC) flow.
Time Frame: Within 12 hours of life
Population: The echocardiograms were not performed on all patients because of lack of available staff
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | Monitored Arm | Control Arm
Number analyzed (Participants) | 16 | 15
ml/kg/min | 83.7 (43.1) | 92.2 (42.3)

ADVERSE EVENTS:
Arm/Group | Monitored Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 3/24 | 1/24
Serious Adverse Events (participants affected / at risk) | 2/24 | 1/24
Other Adverse Events (participants affected / at risk) | 2/24 | 2/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Monitored Arm (N=24) | Control Arm (N=24)
Severe IVH or PVL (Nervous system disorders) | 2 (2) | 1 (1) — severe intracranial hemorrhage or Periventricular Leukomalacia
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Monitored Arm (N=24) | Control Arm (N=24)
air leak (Respiratory, thoracic and mediastinal disorders) | 2 | 2 — an air leak is a pneumothorax

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes